CLINICAL TRIAL: NCT03910738
Title: TOTEM RRMS : TestOsterone TreatmEnt on Neuroprotection and Myelin Repair in Relapsing Remitting Multiple Sclerosis
Acronym: TOTEM-RRMS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Bayer (Industry); Fédération Hospitalo-Universitaire NEUROGENYCS (Unknown); Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7109
Record Dates: First submitted 2019-04-01; First posted 2019-04-10 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Neuroprotection; Remyelination; Relapsing Remitting Multiple sclerosis; Testosterone undecanoate; Diffusion tensor Imaging
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Solutions; Injections; Quality of Life; Exercise

STUDY DESIGN:
Intervention Model Description: multicenter, randomized, parallel-group, double-blind, placebo-controlled phase 2 trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone treatment (Nebido®) (Experimental): "Treatment/Nebido®" arm: in this experimental arm, each patient will be injected intramuscularly with 1000 mg / 4 ml of testosterone undecanoate (Nebido®).
  Treatment will be injected at baseline, week 6, 18, 30, 42 and 54
  Interventions: Drug: Nebido® Testosterone Undecanoate 1000 Mg/4 mL Solution for Injection; Procedure: MRI; Behavioral: Assessment of impact of MS on cognition; quality of life; fatigue; anxiety/depression and work and activities; Behavioral: Assessment of disability
- Placebo (Placebo Comparator): "Placebo" arm: In this arm, each patient will be injected intramuscularly with 4 ml of placebo solution.
  Placebo will be injected at baseline, week 6, 18, 30, 42 and 54
  Interventions: Drug: Placebo 4 mL Solution for Injection; Procedure: MRI; Behavioral: Assessment of impact of MS on cognition; quality of life; fatigue; anxiety/depression and work and activities; Behavioral: Assessment of disability

INTERVENTIONS:
Drug: Nebido® Testosterone Undecanoate 1000 Mg/4 mL Solution for Injection — Active treatment (Nebido® Testosterone Undecanoate ) will be injected at Baseline, at week 6 and then every 12 weeks (Week 18, 30, 42 and 54)
  Arms: Testosterone treatment (Nebido®)
Drug: Placebo 4 mL Solution for Injection — Placebo will be injected at Baseline, at week 6 and then every 12 weeks (Week 18, 30, 42 and 54)
  Arms: Placebo
Procedure: MRI — Conventional MS sequences (OFSEP recommendations) and unconventional MRI sequences (Baseline, week 30 and 66)
Behavioral: Assessment of impact of MS on cognition; quality of life; fatigue; anxiety/depression and work and activities — BICAMS; SF-36 and EQ-5D-3L; MFIS; HADS; WPAI:MS (at baseline, week 30 and 66)
Behavioral: Assessment of disability — EDSS (Baseline, week 30 and 66)

SUMMARY:
Centra nervous system (CNF) damage in multiple sclerosis (MS), are mainly attributed to myelin destruction, axonal abnormalities and subsequent degeneration, and are responsible for serious deficiencies. Current therapies are focused on the treatment of inflammation with several types of anti-inflammatory agents. However, there is an urgent need for innovative therapies promoting neuroregeneration and particularly myelin repair.

It has been demonstrated that testosterone can act through neural androgen receptors to promote proliferation and differentiation of oligodendrocyte precursors into mature oligodendrocytes in a cuprizone-induced animal model of demyelination. The rare clinical trials on testosterone are mainly exploratory. Here, we sought to demonstrate an effect of testosterone supplementation in testosterone-deficient patients in a multicenter, randomized, parallel-group, double-blind, placebo-controlled phase 2 trial.

The main objective will be to determine the neuroprotective and remyelinating effects of testosterone using tensor diffusion imaging techniques and thalamic atrophy analyzes.

As secondary objectives, we would like to study the impact of testosterone supplementation on other conventional and unconventional MRI parameters and on clinical outcomes (cognition, fatigue, quality of life, impact on work / activity and anxiety / depression).

ELIGIBILITY:
Inclusion Criteria:

* Man between 18 and 55 years
* Patient affiliated to a social health insurance plan
* Patient able to understand the objectives and risks related to the research and able to comply with the requirements of the protocol throughout the duration of the study
* Patient having been informed of the results of the prior medical examination
* Patient having signed an informed consent
* Confirmed and documented diagnosis of MS, as defined by the revised McDonald criteria,
* Patient who have been receiving one of the following disease modifying therapies for at least one year prior to randomization: natalizumab , fingolimod, ponesimod, ocrelizumab, or ofatumumab, in accordance with their prescribing information. Switching from one molecule to another during the previous year is also permitted, provided that the switch was motivated by a non-neurological reason (relapse, MRI activity). Patients receiving ocrelizumab within 6 to 9 months are eligible, provided they have received full-dose ocrelizumab for at least 2 years.
* Biological hypogonadism defined by serum total testosterone levels below 20 nmol / L (checked by blood sampling during the screening visit)
* For patients under natalizumab : Negative status for JC virus or JC virus synthesis index ≤ 1.5 (checked by blood sampling at the inclusion visit)
* No relapses in the year prior to inclusion
* Disability status during the selection visit with an EDSS score of 0 to 7 (verified by questionnaire during the inclusion visit)
* Stable neurological state in the month preceding randomization

Exclusion Criteria:

* Patients with progressive MS (primary or secondary)
* Patients with hypogonadism with clinical symptoms and treated with androgens
* Patients with PSA (prostate specific antigen)> 2.5 ng / ml (for an age less than 49 years old) or > 3.5 ng / ml (for age ≥ 50 years) (checked by a blood test at the inclusion visit)
* Patients with a hematocrit level > 54% (checked by blood sampling during the inclusion visit)
* Patients refusing or unable to undergo an MRI
* Patients with any other disease other than MS that may contribute to neurological symptoms and signs or affect their evaluation
* Patients with neurological signs compatible with progressive multifocal leukoencephalopathy (PML) or confirmed leukoencephalopathy
* Patients diagnosed with untreated sleep apnea
* Patients with or having had cancer or tumors of the liver, heart, kidney, prostate or mammary gland
* Patients with cardiovascular, renal, hepatic, hematological, gastrointestinal, pulmonary, uncontrolled diseases
* Patients wishing to procreate during the study period
* Patients with chronic infectious disease
* Patients with organic or psychiatric disease compromise their ability to understand the information given and to follow the protocol
* Patients with a history of hypersensitivity to treatment or any of the excipients, or drugs of similar chemical classes
* Patients who used experimental drugs and / or who participated in clinical drug trials in the 6 months prior to selection
* Patient in exclusion period (determined by previous study or in progress)
* Impossibility of giving information to the patient (subject in emergency situation, difficulties in understanding the subject or other)
* Incapacitated subject (subject to a legal protection measure: safeguard of justice, curatorship, guardianship, future protection mandate, family habilitation)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — male
Enrollment: 40 (Estimated)
Dates: Start 2019-10-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change on MRI binary criterion combining thalamic atrophy and modification in transverse diffusivity of lesions | At baseline, week 30 and week 66 (end of study)
  The primary endpoint is a binary criterion comparing the success rate in each treatment group, defined by thalamic atrophy lower than 0.5% and modification in transverse diffusivity of lesions lower than 0.5% per year compared between baseline and week 66 in each group.

SECONDARY OUTCOMES:
Evolution of the number of T1 hypointense lesions as detected by conventional MRI | At baseline, week 30 and week 66 (end of study)
  Efficacy will be assessed by comparing results between the 2 groups and in each group between baseline, week 30 and week 66.
Evolution of the volume of T1 hypointense lesions as detected by conventional MRIconventional MRI | At baseline, week 30 and week 66 (end of study)
  Efficacy will be assessed by comparing results between the 2 groups and in each group between baseline, week 30 and week 66.
Evolution of the number of new or enlarged T2 lesions as detected by conventional MRI | At baseline, week 30 and week 66 (end of study)
  Efficacy will be assessed by comparing results between the 2 groups and in each group between baseline, week 30 and week 66.
Evolution of the volume of new or enlarged T2 lesions as detected by conventional MRI | At baseline, week 30 and week 66 (end of study)
  Efficacy will be assessed by comparing results between the 2 groups and in each group between baseline, week 30 and week 66.
Evolution of the total volume of hyper-intensity FLAIR lesion as detected by conventional MRI | At baseline, week 30 and week 66 (end of study)
  Efficacy will be assessed by comparing results between the 2 groups and in each group between baseline, week 30 and week 66.
Evolution of diffusion tensor imaging (NODDI) as detected by unconventional MRI | At baseline, week 30 and week 66 (end of study)
  Efficacy will be assessed by comparing results between the 2 groups and in each group between baseline, week 30 and week 66.
Evolution of quantitative magnetization transfer imaging (MPF) as detected by unconventional MRI | At baseline, week 30 and week 66 (end of study)
  Efficacy will be assessed by comparing results between the 2 groups and in each group between baseline, week 30 and week 66.
Evolution of cognitive performance as measured by Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) | At baseline, week 30 and week 66 (end of study)
  BICAMS is a composite cognitive assessment tool comprising of the three components: Symbol Digit Modalities Test (SDMT), California Verbal Learning Test-II (CVLT-II) and Brief visuospatial memory test- Revised (BVMT-R). Efficacy will be assessed by comparing the composite score between the 2 groups and in each group between baseline, week 30 and week 66.
Changes in quality of life as measured by the SF-36 questionnaire | At baseline, week 30 and week 66 (end of study)
  SF-36 questionnaire is a 36-item Short Form survey designed to examine the perceived health status measured in eight health concepts. Answers to each question are scored and summed to produce raw scale scores for each health concept. Efficacy will be assessed by comparing scores between the 2 groups and in each group between baseline, week 30 and week 66.
Changes in quality of life related to health as measured by the EQ-5D-3L (European Quality of Life in 3 Dimensions) questionnaire. | At baseline, week 30 and week 66 (end of study)
  EQ-5D-3L is a standardized instrument used as a measure of health outcome. It is a health questionnaire that consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. Efficacy will be assessed by comparing the composite scores between the 2 groups and in each group between baseline, week 30 and week 66.
Changes in work productivity and daily activities due to MS, as assessed by the WPAI:MS questionnaire (Work Productivity and Activity Impairment in MS). | At baseline, week 30 and week 66 (end of study)
  WPAI questionnaire measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (work time missed) 2. Presenteeism (impairment at work / reduced on-the-job effectiveness) 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism) 4. Activity Impairment. WPAI outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity. Efficacy will be assessed by comparing score between the 2 groups and in each group between baseline, week 30 and week 66.
Changes in fatigue, measured by the Multidimensional Fatigue Impact Scale (MFIS) | At baseline, week 30 and week 66 (end of study)
  MFIS is a 21-item questionnaire that assesses overall self-reported fatigue. Subjects rate agreement with a series of statements on a scale of 0 (rarely) to 4 (almost always), in context of their fatigue over the preceding four weeks. Total possible score of 84. Individuals with an MFIS score of > 38 are considered to experience moderate to severe "fatigue". Efficacy will be assessed by comparing score between the 2 groups and in each group between baseline, week 30 and week 66.
Changes in anxiety and depression as measured by the Hospital assessment for Anxiety and Depression Scale (HADS) questionnaire | At baseline, week 30 and week 66 (end of study)
  HADS is a 14-item self-rating scale that assesses anxiety and depression. Each question is scored on a scale ranging from 0 to 3. Responses are summed to provide separate scores for anxiety and depression that range from 0 to 21. For each corresponding subscale, a total score of 0-7 equals normal, 8-10 equals borderline case, and 11-21 equals case. Efficacy will be assessed by comparing score between the 2 groups and in each group between baseline, week 30 and week 66.
Evolution of disability measured MS specific Expanded Disability Status scale (EDSS) | At baseline, week 30 and week 66 (end of study)
  EDSS measures disability status on a scale ranging from 0 to 10, in eight functional system scale: motor, sensory, cerebellar, brain stem, visual, mental, sphincter and other systems. The EDSS is formed on the score in each functional system; higher scores indicating more disability (0 = normal examination and 10= death from MS). Efficacy will be assessed by comparing score between the 2 groups and in each group between baseline, week 30 and week 66.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From Visit 0/baseline to end of study visit (66 weeks)
  Safety of treatment will be followed by the number and type of adverse or severe adverse events (AE/SAE) throughout the protocol (from baseline to week 66)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent D KREMER, MD, Principal Investigator — CHU Strasbourg
Locations (5):
- France (5):
  - CHU de Besançon, Besançon
  - CHU Nancy, Nancy
  - Hôpital Pitié-Salpêtrière, Paris
  - CHU de Rennes/Pontchaillou, Rennes
  - CHRU de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Metzger-Peter K, Kremer LD, Edan G, Loureiro De Sousa P, Lamy J, Bagnard D, Mensah-Nyagan AG, Tricard T, Mathey G, Debouverie M, Berger E, Kerbrat A, Meyer N, De Seze J, Collongues N. The TOTEM RRMS (Testosterone Treatment on neuroprotection and Myelin Repair in Relapsing Remitting Multiple Sclerosis) trial: study protocol for a randomized, double-blind, placebo-controlled trial. Trials. 2020 Jun 29;21(1):591. doi: 10.1186/s13063-020-04517-6. PMID 32600454